CLINICAL TRIAL: NCT04290871
Title: Nitric Oxide Gas Inhalation Therapy for Severe Acute Respiratory Syndrome Due to COVID-19.
Brief Title: Nitric Oxide Gas Inhalation for Severe Acute Respiratory Syndrome in COVID-19.
Acronym: NOSARSCOVID
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study will start to enroll patients soon
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NO-SARS-COVID-19
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronavirus Covid-19 Infection Variant Omicron; SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Nitric Oxide gas will be administered in the ventilatory circuit.
  Interventions: Drug: Nitric Oxide Gas
- Control Group (Sham Comparator): The delivery system will be set up anyway without study gas administration
  Interventions: Other: The delivery system will be set up anyway without study gas administration

INTERVENTIONS:
Drug: Nitric Oxide Gas — Inspired NO/N2 will be delivered at 80 parts per million (ppm) in the first 48 hours of enrollment (within 48 hours after initiation of mechanical ventilation). Weaning from NO will start after 48-h consecutive NO inhalation. The physicians will follow their own institutional weaning protocols.
  Other Names: Nitric Oxide inhalation
  Arms: Treatment Group
Other: The delivery system will be set up anyway without study gas administration — The delivery system will be set up anyway without study gas administration
  Arms: Control Group

SUMMARY:
The investigators will enroll 104 patients with severe COVID-19 infection that mechanical ventilation is needed for respiratory support. Patients will be randomized to receive either inhaled nitric oxide (per protocol) or a placebo. ICU Standards of care will be the institution's own protocols (such as ventilation strategies and use and dose of antivirals and antimicrobials, steroids, inotropic and vasopressor agents).

DETAILED DESCRIPTION:
The outbreak of COVID-19 and its global pandemic have posed a threat to public health. The deadly virus, SARS-CoV-2, has been evolving to new, more infectious variant and other lineages with additional immune escape mutations. The highly transmissible Omicron variant has been present for around one year and has supplanted Delta as the leading strain in the global pandemic. Although the severity of symptoms caused by the Omicron variant is significantly reduced when compared to its earlier variants, people who are infected with Omicron have the full spectrum of disease, everything from asymptomatic infection all the way through severe disease and death. People with underlying conditions, advanced age, and unvaccinated can have a severe form of COVID-19 following infection from Omicron. On December 7, 2022, the State Council of China issued an announcement on further optimization of measures for preventing and controlling the COVID-19 epidemic ( easing of rigorous "zero COVID" policies). Since then, the rapid spread of COVID-19 has caused surge of COVID-19 infections in majority of China, which caused a dramatic increase of severe cases.

In severe cases with COVID-19 infection significantly affects the respiratory functions by massively disrupting the pulmonary oxygenation and activating the synthesis of proinflammatory cytokines, inducing severe oxidative stress, enhanced vascular permeability, and endothelial dysfunction which have rendered researchers and clinicians to depend on prophylactic treatment due to the unavailability of proper disease management approaches. Inhaled nitric oxide gas (NO) has shown antiviral activity against Coronavirus during the 2003 SARS outbreak. Previous studies have indicated that nitric oxide (NO) application appears to be significant concerning the antiviral activities, antioxidant, and anti-inflammatory properties in relieving disease-related symptoms. Inhaled nitric oxide had been widely used during the Covid-19 pandemic. In the scoping and systemic reviews, it was demonstrated that nitric oxide inhalation was effective in improve oxygenation, cardiopulmonary function, and fasten virus clearance. The investigators designed this study to assess whether inhaled NO improves respiratory recovery in patients affected with severe COVID-19 infection.

Here, the investigators propose a randomized clinical trial aimed to improve recovery of the disease in patients with severe acute respiratory syndrome.

Control group: the institutional standard of care will be delivered. Treatment group: In addition to standard therapy, the subjects will receive inhalation of NO. Inspired NO/N2 will be delivered at 80 parts per million (ppm) in the first 48 hours of enrollment (within 48 hours after initiation of mechanical ventilation). Weaning from NO will start after 48-h consecutive NO inhalation. Physician will follow their own institutional weaning protocols. In the absence of institutional protocols, NO will be reduced every 4 hours in step-wise fashion starting from 40 ppm to 20, 10, 5, 3, 2 and 1 ppm. If hypoxemia (SpO2 < 93%) or acute hypotension (systolic blood pressure < 90 mmHg) occurs during weaning, NO should be increased to a prior higher concentration.

Safety: prolonged treatment with inhaled NO can lead to increased methemoglobin levels. Blood levels of methemoglobin will be monitored via a non-invasive CO-oximeter or MetHb levels in blood. If methemoglobin levels rise above 5% at any point of the study, inhaled NO concentration will be halved.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed Covid-19 infection
3. Severe cases of Covid-19 infection needs mechanical ventilation

Exclusion Criteria:

1. Physician makes a decision that trial involvement is not in the patient's best interest or any condition that does not allow the protocol to be followed safely
2. Pregnant or positive pregnancy test in a pre-dose examination
3. mechanical ventilation initiated for more than 48 hrs
4. Rescue Use ECMO
5. With severe organ dysfunction or failure (Child Pugh≥12, eGFRC30 ml/min/1.73m2, on RRT or dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-16 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation free days (VFDs) | 28 days since beginning of treatment
  count the days that patients do not need mechanical ventilation

SECONDARY OUTCOMES:
Survival at 28 days | 28 days
  count the number of patients that survive to 28 days after randomization
Survival at 90 days | 90 days
  count the number of patients that survive to 90 days after randomization
WHO COVID Ordinal Outcomes Scale | 28 days
  8 score scale, where no limitation of activity =1, death = 8
time to improvement of oxygenation | through oxygenation improvement, an average of 2 days
  time from randomization to PaO2/FiO2 ≥300 at room air
MODS needs life support | 28 days
  Incidence of organ failure need support of RRT, VA-ECMO, LVAD, IABP, Prone ventilation, etc
duration of mechanical ventilation | through wean of mechanical ventilation, an average of 10 days
  days when mechanical ventilation are used
Length of ICU stay and hospital stay | through discharge from ICU or hospital, an average of 20 days
  count days when patients stay in ICU and hospital
SOFA score | at 48 hours, 72 hours, and 7 days after randomization
  Sequential (sepsis-related) organ failure assessment (SOFA) score.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, MD, PhD, Principal Investigator — Air Force Military Medical University, China; Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Chen L, Liu P, Gao H, Sun B, Chao D, Wang F, Zhu Y, Hedenstierna G, Wang CG. Inhalation of nitric oxide in the treatment of severe acute respiratory syndrome: a rescue trial in Beijing. Clin Infect Dis. 2004 Nov 15;39(10):1531-5. doi: 10.1086/425357. Epub 2004 Oct 22. PMID 15546092
- [Background] Keyaerts E, Vijgen L, Chen L, Maes P, Hedenstierna G, Van Ranst M. Inhibition of SARS-coronavirus infection in vitro by S-nitroso-N-acetylpenicillamine, a nitric oxide donor compound. Int J Infect Dis. 2004 Jul;8(4):223-6. doi: 10.1016/j.ijid.2004.04.012. PMID 15234326
- [Background] Valsecchi C, Winterton D, Safaee Fakhr B, Collier AY, Nozari A, Ortoleva J, Mukerji S, Gibson LE, Carroll RW, Shaefi S, Pinciroli R, La Vita C, Ackman JB, Hohmann E, Arora P, Barth WH Jr, Kaimal A, Ichinose F, Berra L; DELiverly oF iNO (DELFiNO) Network Collaborators. High-Dose Inhaled Nitric Oxide for the Treatment of Spontaneously Breathing Pregnant Patients With Severe Coronavirus Disease 2019 (COVID-19) Pneumonia. Obstet Gynecol. 2022 Aug 1;140(2):195-203. doi: 10.1097/AOG.0000000000004847. Epub 2022 Jul 6. PMID 35852269
- [Background] Fang W, Jiang J, Su L, Shu T, Liu H, Lai S, Ghiladi RA, Wang J. The role of NO in COVID-19 and potential therapeutic strategies. Free Radic Biol Med. 2021 Feb 1;163:153-162. doi: 10.1016/j.freeradbiomed.2020.12.008. Epub 2020 Dec 22. PMID 33347987
- [Background] Garfield B, McFadyen C, Briar C, Bleakley C, Vlachou A, Baldwin M, Lees N, Price S, Ledot S, McCabe C, Wort SJ, Patel BV, Price LC. Potential for personalised application of inhaled nitric oxide in COVID-19 pneumonia. Br J Anaesth. 2021 Feb;126(2):e72-e75. doi: 10.1016/j.bja.2020.11.006. Epub 2020 Nov 14. No abstract available. PMID 33288208
- [Background] Montiel V, Lobysheva I, Gerard L, Vermeersch M, Perez-Morga D, Castelein T, Mesland JB, Hantson P, Collienne C, Gruson D, van Dievoet MA, Persu A, Beauloye C, Dechamps M, Belkhir L, Robert A, Derive M, Laterre PF, Danser AHJ, Wittebole X, Balligand JL. Oxidative stress-induced endothelial dysfunction and decreased vascular nitric oxide in COVID-19 patients. EBioMedicine. 2022 Mar;77:103893. doi: 10.1016/j.ebiom.2022.103893. Epub 2022 Feb 23. PMID 35219085
- [Background] Ghosh A, Joseph B, Anil S. Nitric Oxide in the Management of Respiratory Consequences in COVID-19: A Scoping Review of a Different Treatment Approach. Cureus. 2022 Apr 5;14(4):e23852. doi: 10.7759/cureus.23852. eCollection 2022 Apr. PMID 35530860
- [Result] Al Sulaiman K, Korayem GB, Altebainawi AF, Al Harbi S, Alissa A, Alharthi A, Kensara R, Alfahed A, Vishwakarma R, Al Haji H, Almohaimid N, Al Zumai O, Alrubayan F, Asiri A, Alkahtani N, Alolayan A, Alsohimi S, Melibari N, Almagthali A, Aljahdali S, Alenazi AA, Alsaeedi AS, Al Ghamdi G, Al Faris O, Alqahtani J, Al Qahtani J, Alshammari KA, Alshammari KI, Aljuhani O. Evaluation of inhaled nitric oxide (iNO) treatment for moderate-to-severe ARDS in critically ill patients with COVID-19: a multicenter cohort study. Crit Care. 2022 Oct 3;26(1):304. doi: 10.1186/s13054-022-04158-y. PMID 36192801